CLINICAL TRIAL: NCT02096445
Title: Neurocognitive Robot-assisted Rehabilitation of Hand Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roger Gassert (Other)
Responsible Party: Sponsor-Investigator, Roger Gassert, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIV-13-02-009921; 2013-MD-0002 (Other: Swissmedic)
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: stroke; acute; rehabilitation; robot therapy; hand function; fine motor skills; neurocognitive; sensory; Perfetti; haptics
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot group (Experimental): Receive robot-assisted neurocognitive therapy instead of conventional neurocognitive therapy.
  (4 x 45 min/week)
  Interventions: Device: robot-assisted neurocognitive therapy of hand function
- Control group (Active Comparator): Receive dose-matched conventional neurocognitive therapy
  Interventions: Other: Conventional neurocognitive rehabilitation

INTERVENTIONS:
Device: robot-assisted neurocognitive therapy of hand function — 2 degrees-of-freedom hand rehabilitation robot to train fine motor skills during grasping and forearm rotation.
  Other Names: Rehabilitation robot ReHapticKnob
  Arms: Robot group
Other: Conventional neurocognitive rehabilitation — Use sensory perception (tactile, proprioception but not vision!) to solve a by the therapist guided (passive) or patient controlled (active) therapy task, e.g. discrimination/identification of different spring resistances, sponges, different sized blocks, etc.
  Other Names: Perfetti-concept
  Arms: Control group

SUMMARY:
The aim of this project is to clinically evaluate a novel robot-assisted therapeutic approach to train sensorimotor hand function after stroke. It combines the profound experience of the clinic Hildebrand in neurocognitive therapy - involving brain and mind in the task and training both the motor and the sensory system - with the advanced haptic robotic technology of the Rehabilitation Engineering Lab at the Swiss Federal Institute of Technology Zurich (ETH Zurich), allowing unmet interaction with the hand through the simulation of virtual objects with various mechanical properties. In a randomized controlled clinical trial, 10 sub-acute stroke patients will receive four weeks of robotic therapy sessions, integrated seamlessly into their daily rehabilitation program, while 10 other patients will receive conventional therapy. The investigators will assess baseline performance in an initial clinical and robotic assessment, with another assessment at the end of the four-week period, and in follow-ups four weeks and six months later. The contents of the patient-tailored robotic therapy sessions will match those of the conventional therapy as closely as possible. This study will demonstrate the feasibility of including robotic therapy of hand function into the daily rehabilitation program, and investigate the acceptance from patients and therapists. The investigators expect increased training intensity during the robotic therapy session compared to conventional sessions with similar contents, as well as novel insights into the recovery process of both the motor and the sensory system during the four weeks of therapy, through advanced robotic assessments integrated into the training sessions. This project is a first step towards making such robotic therapy available to patients as integration into the conventional individual therapy program (e.g. for self-training), and towards transferring this technology to the home environment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-90 years old
* hemisyndrome (central paralysis of the upper extremity, and all degrees of weakness: M0 - M5 on the paresis scale) as a result of a first stroke
* sub-acute lesion not more than 6 weeks post ictus

Exclusion Criteria:

* insufficient state of consciousness
* severe aphasia
* severe cognitive deficits
* severe pathologies of the upper extremity of traumatic or rheumatic nature
* severe pain in the affected arm
* Patients with pacemakers and other active implants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Motor impairment of the upper limb | Change from Baseline in motor impairment of the upper limb at 4 weeks
  Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale of the upper limb (total of 66 points)

SECONDARY OUTCOMES:
Motor impairment of the upper limb | Change from Baseline in motor impairment of the upper limb at 8 weeks
  Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale of the upper limb (total of 66 points)
Motor impairment of the upper limb | Change from Baseline in motor impairment of the upper limb at 6 months
  Motor impairment of the upper limb is measured by the means of the Fugl-Meyer Assessment Scale of the upper limb (total of 66 points)
Functional improvement in dexterity | Change from Baseline in functional improvement of dexterity of the upper limb at 4 weeks
  Functional improvement in dexterity is assessed with the Box and Block Test
Functional improvement in dexterity | Change from Baseline in functional improvement of dexterity of the upper limb at 8 weeks
  Functional improvement in dexterity is assessed with the Box and Block Test
Functional improvement in dexterity | Change from Baseline in functional improvement of dexterity of the upper limb at 6 months
  Functional improvement in dexterity is assessed with the Box and Block Test
Spasticity level of the upper limb | Change from Baseline in spasticity level of the upper limb at 4 weeks
  Spasticity level is measured with the Modified Ashworth Scale
Spasticity level of the upper limb | Change from Baseline in spasticity level of the upper limb at 8 weeks
  Spasticity level is measured with the Modified Ashworth Scale
Spasticity level of the upper limb | Change from Baseline in spasticity level of the upper limb at 6 months
  Spasticity level is measured with the Modified Ashworth Scale
Tactile and proprioceptive sensory function of the upper limb | Change from Baseline in Tactile and proprioceptive sensory function of the upper limb at 4 weeks
  Tactile and proprioceptive sensory function of the upper limb is assessed with the Erasmus MC (Medical Center) Nottingham Sensory Assessment
Tactile and proprioceptive sensory function of the upper limb | Change from Baseline in tactile and proprioceptive sensory function of the upper limb at 8 weeks
  Tactile and proprioceptive sensory function of the upper limb is assessed with the Erasmus MC Nottingham Sensory Assessment
Tactile and proprioceptive sensory function of the upper limb | Change from Baseline in tactile and proprioceptive sensory function of the upper limb at 6 months
  Tactile and proprioceptive sensory function of the upper limb is assessed with the Erasmus MC Nottingham Sensory Assessment
Neglect | Change from Baseline in neglect at 4 weeks
  Neglect is assessed with the Albert's test of neglect
Neglect | Change from Baseline in neglect at 8 weeks
  Neglect is assessed with the Albert's test of neglect
Neglect | Change from Baseline in neglect at 6 months
  Neglect is assessed with the Albert's test of neglect
Cognitive impairment | Change from Baseline in cognitive impairment at 4 weeks
  Cognitive impairment is assessed with the Mini Mental State Examination
Cognitive impairment | Change from Baseline in cognitive impairment at 8 weeks
  Cognitive impairment is assessed with the Mini Mental State Examination
Cognitive impairment | Change from Baseline in cognitive impairment at 6 months
  Cognitive impairment is assessed with the Mini Mental State Examination
Frontal lobe function | Change from Baseline in frontal lobe function at 4 weeks
  Frontal lobe function is assessed with the Frontal assessment battery
Frontal lobe function | Change from Baseline in frontal lobe function at 8 weeks
  Frontal lobe function is assessed with the Frontal assessment battery
Frontal lobe function | Change from Baseline in frontal lobe function at 6 months
  Frontal lobe function is assessed with the Frontal assessment battery
Aphasia | Change from Baseline in aphasia at 4 weeks
  Aphasia is assessed with the Aachener Aphasia Test
Aphasia | Change from Baseline in aphasia at 8 weeks
  Aphasia is assessed with the Aachener Aphasia Test
Aphasia | Change from Baseline in aphasia at 6 months
  Aphasia is assessed with the Aachener Aphasia Test
Attention | Change from Baseline in attention at 4 weeks
  Attention is assessed with the test to identify attention
Attention | Change from Baseline in attention at 8 weeks
  Attention is assessed with the test to identify attention
Attention | Change from Baseline in attention at 6 months
  Attention is assessed with the test to identify attention

CONTACTS AND LOCATIONS:
Overall Officials: Roger Gassert, Prof. Dr., Study Director — Rehabilitation Engineering Lab, ETH Zurich
Locations (1):
- Clinica Hildebrand Centro di riabilitazione Brissago, Brissago, Canton Ticino, Switzerland

REFERENCES:
- [Result] Metzger JC, Lambercy O, Califfi A, Conti FM, Gassert R. Neurocognitive robot-assisted therapy of hand function. IEEE Trans Haptics. 2014 Apr-Jun;7(2):140-9. doi: 10.1109/TOH.2013.72. PMID 24968378
- [Derived] Ranzani R, Lambercy O, Metzger JC, Califfi A, Regazzi S, Dinacci D, Petrillo C, Rossi P, Conti FM, Gassert R. Neurocognitive robot-assisted rehabilitation of hand function: a randomized control trial on motor recovery in subacute stroke. J Neuroeng Rehabil. 2020 Aug 24;17(1):115. doi: 10.1186/s12984-020-00746-7. PMID 32831097
- [Derived] Metzger JC, Lambercy O, Califfi A, Dinacci D, Petrillo C, Rossi P, Conti FM, Gassert R. Assessment-driven selection and adaptation of exercise difficulty in robot-assisted therapy: a pilot study with a hand rehabilitation robot. J Neuroeng Rehabil. 2014 Nov 15;11:154. doi: 10.1186/1743-0003-11-154. PMID 25399249
- See also: Homepage of the investigator's laboratory — http://www.relab.ethz.ch